CLINICAL TRIAL: NCT02660086
Title: Promoting Employee Health Through The Worksite Food Environment
Acronym: ChooseWell 365
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01HL125486 (NIH); R01DK114735 (NIH)
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Weight; Food Choice; Nutrition Intake
Keywords: Weight; Prevention; Food choice; Nutrition; Behavior change; Behavioral economics; Feedback; Incentives
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized feedback (Experimental): Emails and letters providing personalized nutrition feedback about food choices and health, social norms, and financial incentives for healthy food choices
  Interventions: Behavioral: Personalized nutrition feedback
- Control (No Intervention): Monthly letters with general nutrition information

INTERVENTIONS:
Behavioral: Personalized nutrition feedback — Automated personalized nutrition feedback about cafeteria food purchases (weekly); social norms and small financial incentives to promote healthy purchases (monthly)
  Arms: Personalized feedback

SUMMARY:
This project tests a scalable and sustainable approach to weight gain prevention in a population of employees by using the worksite environment to deliver personalized feedback about worksite food purchases, daily calorie goals, social norms for healthy eating, and financial incentives for healthy food purchases. In the future, similar strategies could be adopted by other worksites, institutions, and food retailers and could contribute to the long-term environmental and social changes needed to reverse the obesity epidemic in the United States and worldwide.

The overall objective of ancillary studies added on to this project is to examine the psychological traits, cognitive skills, and genes that may influence the impact of the behavioral intervention to promote healthy diet and weight among employees at a large hospital worksite.

DETAILED DESCRIPTION:
Adults in the United States gain an average of 1-2 pounds a year. Interventions to prevent weight gain at the population level are needed to reverse the rising prevalence of obesity. Although individual-level interventions can result in large weight changes among small groups of individuals, achieving changes in the population will require long-term strategies that create healthier food environments, establish new social norms, and improve motivation and skills for healthy lifestyle behaviors. The worksite is ideal for interventions to address weight and lifestyle behaviors because a majority of adults are employed, and provisions in the Affordable Care Act encourage worksite wellness. Our research team at Massachusetts General Hospital (MGH) has demonstrated that behavioral economics strategies, including traffic-light labels, choice architecture, social norms, and financial incentives, improve employees' healthy food choices. The proposed project will address the critical next phase of this research to determine if a worksite intervention delivered through the food environment can prevent weight gain and reduce cardiovascular risk of employees. This project builds on the established traffic-light labeling system at MGH and tests an intervention that aims to increase nutrition knowledge, motivate change in lifestyle behaviors, and promote socially normative behavior for healthier lifestyles among employees. The intervention will be integrated into the flow of the work day, thus lowering burden to employees and the employer. Study Design: In a randomized controlled trial, 600 MGH employees will be assigned to: 1) an intervention arm with automated, personalized feedback about (a) worksite food purchases and calorie and physical activity goals (weekly emails) and (b) social norm feedback plus small financial incentives for healthy food purchases (monthly letters) or 2) a control arm (standardized monthly letters). Study outcomes will be assessed at 1 year (end of intervention) and 2 year follow-up. The primary outcome is change in weight at 1 year. Secondary outcomes are cardiovascular risk factors, worksite food purchases, and dietary intake (as measured by the Healthy Eating Index). A novel exploratory outcome will be healthy food purchases of co-workers who are socially connected to study subjects. Aim 1 is to determine if employees assigned to the intervention have less weight gain and lower cardiovascular risk factors than the control group at 1 year and 2-year follow-up. Aim 2 is to determine if employees assigned to the intervention group make healthier food choices than the control group at 1 year and 2-year follow-up. Exploratory Aim 3 is to determine if employees socially connected to the intervention group make healthier worksite food choices over 1 year than employees connected to the control group. Implications: This innovative strategy utilizing personalized feedback, social norms, and financial incentives will provide a scalable and sustainable model that could be adopted in other worksite, institutional, and retail settings to prevent obesity at the population level.

The overall objective of the ancillary studies added on to this project is to examine the psychological traits, cognitive skills, and genes that may influence the impact of a behaviorally-informed intervention on dietary choices, weight, and other objective health indicators. This research will expand on the randomized trial by examining psychological traits (impulsivity, self-control, social acceptance), cognitive skills (numeracy, health literacy), and genes (97 known BMI loci) that are associated with obesity and poor health and are specifically targeted by the intervention. We will use validated measures to assess traits and skills and well-established methods for genotyping and calculating genetic risk scores. Aim 1 will determine if psychological traits moderate the behavioral intervention effects on diet and weight. Aim 2 will determine if cognitive skills moderate the behavioral intervention effects on diet and weight. Aim 3 will determine if genetic risk for obesity moderates the intervention effect on weight. In secondary analyses, potential mediators of diet and weight outcomes, including dietary intent, self-efficacy, reward sensitivity, perceived norms, and perceived stress, will be assessed. Implications: Results of this research will l will inform the future design and implementation of more effective, tailored, and sustainable population approaches for obesity prevention.

ELIGIBILITY:
Inclusion Criteria:

* Employee at Massachusetts General Hospital; uses hospital cafeterias at least 4 times a week and willing to pay for purchases with employee debit card.

Exclusion Criteria:

* Planning to leave employment at MGH in the next year; currently pregnant; currently participating in the MGH employee wellness program Be Fit

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dashti HS, Alimenti K, Levy DE, Hivert MF, McCurley JL, Saxena R, Thorndike AN. Chronotype Polygenic Score and the Timing and Quality of Workplace Cafeteria Purchases: Secondary Analysis of the ChooseWell 365 Randomized Controlled Trial. Curr Dev Nutr. 2023 Feb 18;7(3):100048. doi: 10.1016/j.cdnut.2023.100048. eCollection 2023 Mar. PMID 37181927
- [Derived] McCurley JL, Buckholtz JW, Roberto CA, Levy DE, Anderson EM, Chang Y, Thorndike AN. The association of impulsivity with effects of the ChooseWell 365 workplace nudge intervention on diet and weight. Transl Behav Med. 2023 May 13;13(5):281-288. doi: 10.1093/tbm/ibac103. PMID 36548448
- [Derived] Thorndike AN, McCurley JL, Gelsomin ED, Anderson E, Chang Y, Porneala B, Johnson C, Rimm EB, Levy DE. Automated Behavioral Workplace Intervention to Prevent Weight Gain and Improve Diet: The ChooseWell 365 Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2112528. doi: 10.1001/jamanetworkopen.2021.12528. PMID 34097048
- [Derived] Dashti HS, Hivert MF, Levy DE, McCurley JL, Saxena R, Thorndike AN. Polygenic risk score for obesity and the quality, quantity, and timing of workplace food purchases: A secondary analysis from the ChooseWell 365 randomized trial. PLoS Med. 2020 Jul 21;17(7):e1003219. doi: 10.1371/journal.pmed.1003219. eCollection 2020 Jul. PMID 32692747
- [Derived] Feig EH, Levy DE, McCurley JL, Rimm EB, Anderson EM, Gelsomin ED, Thorndike AN. Association of work-related and leisure-time physical activity with workplace food purchases, dietary quality, and health of hospital employees. BMC Public Health. 2019 Nov 27;19(1):1583. doi: 10.1186/s12889-019-7944-1. PMID 31775714
- [Derived] Levy DE, Gelsomin ED, Rimm EB, Pachucki M, Sanford J, Anderson E, Johnson C, Schutzberg R, Thorndike AN. Design of ChooseWell 365: Randomized controlled trial of an automated, personalized worksite intervention to promote healthy food choices and prevent weight gain. Contemp Clin Trials. 2018 Dec;75:78-86. doi: 10.1016/j.cct.2018.11.004. Epub 2018 Nov 7. PMID 30414448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study- 12-month
Arm/Group | Personalized Feedback | Control
Started | 299 | 303
Completed | 273 | 274
Not Completed | 26 | 29
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Left full-time employment | 12 | 20
Not completed — Missed 12-month follow-up visit | 8 | 4
Not completed — Became ineligible: new job in cafeteria | 1 | 0
Period: Overall Study: 24-month Follow-up
Arm/Group | Personalized Feedback | Control
Started | 281 | 278
Completed | 255 | 254
Not Completed | 26 | 24
Not completed — Left employment after 12 months | 17 | 8
Not completed — Missed 24-month follow-up | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Feedback | Control | Total
Number analyzed (Participants) | 299 | 303 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.0) | 43.8 (12.5) | 43.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 248 | 478
  Male | 69 | 55 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 34
  Not Hispanic or Latino | 282 | 286 | 568
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 246 | 242 | 488
  Black | 28 | 26 | 54
  Asian | 14 | 13 | 27
  Other race or not reported | 11 | 22 | 33
Region of Enrollment [Number; unit: participants]
  United States | 299 | 303 | 602
Education [Count of Participants; unit: Participants]
  High school or some college | 36 | 39 | 75
  College degree | 123 | 117 | 240
  Graduate degree | 138 | 146 | 284
  Not reported | 2 | 1 | 3
Job category [Count of Participants; unit: Participants]
  Administrative or service | 36 | 48 | 84
  Crafts or technicians | 36 | 31 | 67
  Management or professionals | 193 | 184 | 377
  Physicians or PhDs | 34 | 40 | 74
Weight [Mean (Standard Deviation); unit: kg] | 79.8 (18.8) | 77.0 (18.3) | 78.4 (18.6)
Weight category [Count of Participants; unit: Participants]
  Normal weight (BMI <25) | 109 | 119 | 228
  Overweight (BMI 25-29.9) | 92 | 100 | 192
  Obese (BMI >=30) | 98 | 84 | 182
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.6 (6.6) | 27.9 (6.4) | 28.3 (6.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 121.4 (14.4) | 120.4 (14.7) | 120.9 (14.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 71.3 (9.9) | 70.2 (9.9) | 70.7 (9.9)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 183.8 (34.8) | 182.7 (38.2) | 183.2 (36.5)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 102.1 (30.6) | 101.5 (33.2) | 101.8 (31.9)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 63.0 (18.5) | 62.1 (17.4) | 62.5 (17.9)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 94.5 (56.3) | 94.5 (67.0) | 94.5 (61.9)
Hemoglobin A1C [Mean (Standard Deviation); unit: percent] | 5.5 (0.5) | 5.5 (0.6) | 5.5 (0.6)
Percentage green-labeled (healthy) food purchased [Mean (Standard Deviation); unit: percent] — Green-labeled food is the healthiest food in the cafeteria and has a main ingredient of either fruit, vegetable, low-fat dairy, or lean protein AND is low in calories and unhealthy fats.
  percent | 50.1 (16.3) | 52.3 (17.1) | 51.2 (16.7)
Percentage yellow-labeled food purchased [Mean (Standard Deviation); unit: percent] — Yellow-labeled food is considered "less healthy" than green-labeled food but healthier than red-labeled food.
  percent | 34.2 (11.8) | 33.1 (11.9) | 33.6 (11.9)
Percentage red-labeled food purchased [Mean (Standard Deviation); unit: percent] — Red-labeled food is the least healthy food in the cafeteria and is high in calories, unhealthy fats (saturated), or both.
  percent | 15.7 (10.8) | 14.6 (10.9) | 15.1 (10.9)
Healthy purchasing score [Mean (Standard Deviation); unit: units on a scale from 0-100] — Overall score of the healthfulness of foods purchased, weighting the proportion of red, yellow, and green foods. To calculate the score, red foods are weighted 0, yellow are weighted 0.5, and green foods are weighted 1.0. Weighted scores are multiplied x 100, and the range is from 0 (least healthy cafeteria purchases, i.e. all red) to 100 (healthiest cafeteria purchases, i.e. all green).
  units on a scale from 0-100 | 67.2 (12.5) | 68.8 (13.1) | 68.0 (12.8)
Healthy Eating Index Score [Mean (Standard Deviation); unit: units on a scale from 0-100] — Healthy Eating Index Score is a measure of overall dietary quality that was calculated from 2 24-hour dietary recalls. The range is from 0 (lowest diet quality) to 100 (highest diet quality).
  units on a scale from 0-100 | 59.7 (12.3) | 61.0 (12.5) | 60.4 (12.4)
Hypertension [Count of Participants; unit: Participants]
  Hypertension | 51 | 49 | 100
  No hypertension | 248 | 254 | 502
Hyperlipidemia [Count of Participants; unit: Participants]
  Hyperlipidemia | 51 | 60 | 111
  No hyperlipidemia | 248 | 243 | 491
Prediabetes or diabetes [Count of Participants; unit: Participants]
  Diabetes or prediabetes | 20 | 25 | 45
  No diabetes or prediabetes | 279 | 278 | 557
Weight goal [Count of Participants; unit: Participants]
  Lose weight | 248 | 255 | 503
  Maintain weight | 51 | 48 | 99
Current smoker [Count of Participants; unit: Participants]
  Current smoker | 8 | 9 | 17
  Non-smoker | 291 | 294 | 585

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Change in weight from baseline to 12 months
Time Frame: 12 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
kg | 0.6 [0.1 to 1.1] | 0.4 [-0.1 to 0.9]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Test type: Superiority; p = 0.70, Mixed Models Analysis; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.6 to 1.0]

2. Secondary Outcome: Weight Change
Description: Change in weight from baseline to 24 months
Time Frame: 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
kg | 1.5 [0.7 to 2.2] | 0.9 [0.2 to 1.6]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Test type: Superiority; p = 0.20, Mixed Models Analysis; Mean Difference (Net) = 0.6, 95% CI 2-sided [-0.3 to 1.4]

3. Secondary Outcome: Change in Blood Pressure
Description: Change from baseline in mean systolic and diastolic blood pressure (BP).
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
mm Hg
  Change in systolic BP from baseline to 12 months | -1.9 [-3.4 to -0.3] | -0.5 [-2.4 to 1.4]
  Change in systolic BP from baseline to 24 months | -0.2 [-1.9 to 1.6] | -1.7 [-3.4 to 0.1]
  Change in diastolic BP from baseline to 12 months | -2.4 [-3.5 to -1.3] | -0.8 [-2.1 to 0.4]
  Change in diastolic BP from baseline to 24 months | -1.7 [-2.8 to -0.6] | -1.8 [-3.0 to -0.6]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in systolic BP at 12 months; Test type: Superiority; p = 0.24, Mixed Models Analysis; Mean Difference (Net) = -1.3, 95% CI 2-sided [-3.6 to 0.9]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in systolic BP at 24 months; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Net) = 1.5, 95% CI 2-sided [-0.7 to 3.7]
Statistical Analysis 3: Comparison: Personalized Feedback vs Control; Change in diastolic BP at 12 months; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.2 to 0.1]
Statistical Analysis 4: Comparison: Personalized Feedback vs Control; Change in diastolic BP at 24 months; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.5 to 1.6]

4. Secondary Outcome: Change in Total Cholesterol
Description: Change from baseline in mean serum total cholesterol.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
mg/dL
  Change from baseline to 12 months | -0.3 [-3.2 to 2.6] | 1.0 [-2.5 to 4.6]
  Change from baseline to 24 months | 2.5 [-0.7 to 5.6] | 0.9 [-3.3 to 5.0]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in total cholesterol at 12 months; Test type: Superiority; p = 0.54, Mixed Models Analysis; Mean Difference (Net) = -1.3, 95% CI 2-sided [-5.6 to 2.9]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in total cholesterol at 24 months; Test type: Superiority; p = 0.53, Mixed Models Analysis; Mean Difference (Net) = 1.6, 95% CI 2-sided [-3.5 to 6.7]

5. Secondary Outcome: Change in LDL Cholesterol
Description: Change from baseline in mean serum LDL.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
mg/dL
  Change from baseline to 12 months | 0.8 [-1.9 to 3.4] | 2.0 [-0.7 to 4.6]
  Change from baseline to 24 months | 4.9 [1.9 to 7.9] | 3.8 [0.3 to 7.2]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in LDL at 12 months; Test type: Superiority; p = 0.51, Mixed Models Analysis; Mean Difference (Net) = -1.2, 95% CI 2-sided [-4.8 to 2.4]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in LDL at 24 months; Test type: Superiority; p = 0.60, Mixed Models Analysis; Mean Difference (Net) = 1.2, 95% CI 2-sided [-3.4 to 5.7]

6. Secondary Outcome: Change in Triglycerides
Description: Change in mean serum triglycerides.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
mg/dL
  Change from baseline to 12 months | -1.1 [-6.3 to 4.0] | 1.8 [-5.7 to 9.2]
  Change from baseline to 24 months | 1.9 [-2.8 to 6.5] | -2.2 [-7.5 to 3.2]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in triglycerides at 12 months; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = -2.9, 95% CI 2-sided [-10.8 to 5.1]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in triglycerides at 24 months; Test type: Superiority; p = 0.29, Mixed Models Analysis; Mean Difference (Net) = 4.0, 95% CI 2-sided [-3.4 to 11.5]

7. Secondary Outcome: Change in HDL Cholesterol
Description: Change in mean serum HDL.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
mg/dL
  Change from baseline to 12 months | -1.5 [-2.6 to -0.4] | -1.3 [-2.9 to 0.4]
  Change from baseline to 24 months | -2.8 [-4.1 to -1.5] | -2.5 [-3.9 to -1.1]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in HDL at 12 months; Test type: Superiority; p = 0.80, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.9 to 1.5]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in HDL at 24 months; Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.9 to 1.3]

8. Secondary Outcome: Change in Hemoglobin A1C
Description: Change in mean serum hemoglobin A1c.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
Percentage
  Change from baseline to 12 months | -0.1 [-0.1 to 0] | -0.1 [-0.2 to 0]
  Change from baseline to 24 months | -0.1 [-0.1 to 0] | -0.1 [-0.2 to -0.1]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in hemoglobin A1C at 12 months; Test type: Superiority; p = 0.62, Mixed Models Analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.1]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in hemoglobin A1C at 24 months; Test type: Superiority; p = 0.40, Mixed Models Analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [0.0 to 0.1]

9. Secondary Outcome: Change in Green-labeled (Healthy) Food Purchases
Description: Change in cafeteria food purchases labeled green.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: percentage of purchases labeled green
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
percentage of purchases labeled green
  Change from baseline to 12 months | 9.4 [8.0 to 10.7] | 2.0 [0.9 to 3.1]
  Change from baseline to 24 months | 5.7 [4.1 to 7.4] | 0.9 [-0.6 to 2.4]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in green labeled purchases during 12 month intervention (months 1-12) compared to baseline 12 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 7.3, 95% CI 2-sided [5.4 to 9.3]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in green-labeled purhases during 12 month follow-up (months 13-24) compared to 12 month baseline; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 4.8, 95% CI 2-sided [2.9 to 6.8]

10. Secondary Outcome: Change in Red-labeled (Unhealthy) Food Purchases
Description: Change in cafeteria food purchases labeled red.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: percentage of purchases labeled red
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
percentage of purchases labeled red
  Change from baseline to 12 months | -4.8 [-5.5 to -4.0] | -0.9 [-1.6 to -0.2]
  Change from baseline to 24 months | -4.1 [-5.0 to -3.2] | -1.0 [-2.0 to 0.1]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in red labeled purchases during 12 month intervention (months 1-12) compared to baseline 12 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.9, 95% CI 2-sided [-5.0 to -2.7]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in red labeled purchases during 12-month follow up (months 13-24) compared to baseline 12 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -3.1, 95% CI 2-sided [-4.3 to -2.0]

11. Secondary Outcome: Change in Healthy Purchasing Score
Description: Change in overall score of the healthfulness of foods purchased, weighting the proportion of red, yellow, and green foods. To calculate the score, red foods are weighted 0, yellow are weighted 0.5, and green foods are weighted 1.0. Weighted scores are multiplied x 100, and the range is from 0 (least healthy cafeteria purchases, i.e. all red) to 100 (healthiest cafeteria purchases, i.e. all green).
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: score on a scale (range 0-100)
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
score on a scale (range 0-100)
  Change from baseline to 12 months | 7.1 [6.1 to 8.0] | 1.5 [0.7 to 2.2]
  Change from baseline to 24 months | 4.9 [3.8 to 6.0] | 0.9 [-0.2 to 2.0]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in healthy purchasing score during 12 month intervention (months 1-12) compared to baseline 12 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 5.6, 95% CI 2-sided [4.2 to 7.0]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in Healthy Purchasing Score during 12 month follow up (months 13-24) compared to baseline 12 months; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 4.0, 95% CI 2-sided [2.6 to 5.3]

12. Secondary Outcome: Change in Healthy Eating Index Score-15
Description: Change in Healthy Eating Index (HEI) scores. Healthy Eating Index Score is a measure of overall dietary quality that was calculated from two 24-hour dietary recalls. The range is from 0 (lowest diet quality) to 100 (highest diet quality) points.
Time Frame: 12 and 24 months
Population: We conducted an intent-to-treat analysis with all missing data imputed for 12 and 24-month outcomes.
Measure: Mean (95% Confidence Interval); unit: score on a scale (range 0-100)
Arm/Group | Personalized Feedback | Control
Number analyzed (Participants) | 299 | 303
score on a scale (range 0-100)
  Change from baseline to 12 months | 1.1 [-0.5 to 2.8] | -0.5 [-2.3 to 1.3]
  Change from baseline to 24 months | 0.6 [-1.1 to 2.4] | -0.9 [-2.7 to 1.0]
Statistical Analysis 1: Comparison: Personalized Feedback vs Control; Change in HEI scores at 12 months; Test type: Superiority; Mean Difference (Net) = 1.8, 95% CI 2-sided [-0.6 to 4.1]
Statistical Analysis 2: Comparison: Personalized Feedback vs Control; Change in HEI scores at 24 months; Test type: Superiority; Mean Difference (Net) = 1.6, 95% CI 2-sided [-0.7 to 3.8]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Personalized Feedback | Control
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/303
Serious Adverse Events (participants affected / at risk) | 0/299 | 0/303
Other Adverse Events (participants affected / at risk) | 0/299 | 0/303

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT02660086/Prot_SAP_000.pdf